CLINICAL TRIAL: NCT02412319
Title: The Efficacy and Safety of the Anti Hepatitis B Placenta Transfer Factor Injection in the Treatment of HBeAg Positive Chronic Hepatitis B, Randomized, Double Blind, Placebo Controlled, Multi Center Clinical Trial
Brief Title: The Clinical Trial of the Anti Hepatitis B Placenta Transfer Factor Injection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shineway Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SW002
Record Dates: First submitted 2015-03-10; First posted 2015-04-09 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: HBeAg Positive Chronic Hepatitis B
Keywords: HBeAg positive chronic hepatitis B; HBeAg serum conversion rate; HBeAg serum disappearance rate; HBeAg and HBsAg titer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Group (Experimental): Anti-HBV Placenta Transfer Factor Injection: 2mg/4ml, intramuscular injection, the 0-24 week, once every other day; week 24-48, 2 times / week; entecavir tablets: 0.5mg/ tablet / time, daily bedtime fasting oral once, treatment course 96 weeks
  Interventions: Drug: Anti-HBV placenta transfer factor injection
- Comparator Group (Placebo Comparator): Physiological saline injection: 2mg/4ml, intramuscular injection,the 0-24 week, once every other day, week 24-48, 2 times / week; entecavir tablets: 0.5mg/ tablet / time, daily bedtime fasting oral once, treatment course 96 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Anti-HBV placenta transfer factor injection — Anti-HBV Placenta Transfer Factor Injection: 2mg/4ml, intramuscular injection, the 0-24 week, once every other day; week 24-48, 2 times / week; entecavir tablets: 0.5mg/ tablet / time, daily bedtime fasting oral once, treatment course 96 weeks
  Arms: Experimental Group
Other: Placebo — Physiological saline injection: 2mg/4ml, intramuscular injection,the 0-24 week, once every other day, week 24-48, 2 times / week; entecavir tablets: 0.5mg/ tablet / time, daily bedtime fasting oral once, treatment course 96 weeks
  Arms: Comparator Group

SUMMARY:
Asses the efficacy and safety of the Anti hepatitis B placenta transfer factor injection in the treatment of HBeAg positive chronic hepatitis B.

DETAILED DESCRIPTION:
This study using entecavir tablets as basic therapy, is a randomized, double-blind, placebo-controlled multi center study, including the screening period (-4 weeks), baseline and treatment period (96 weeks). The treatment period of first 48 weeks, using entecavir tablets as basic treatment, placebo-controlled trials; the second 48 weeks, taking entecavir tablets alone, continue observation experiment.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-65, sex not limited;
2. patients with HBeAg positive chronic hepatitis B: Screening HBsAg positive for more than 6 months; screening HBeAg positive; screening serum HBV DNA≥1.0×105U/ml；
3. 2 * ULN (2 times the upper limit of normal value) < ALT <10 * ULN (10 times the upper limit of normal value);;
4. total bilirubin <51μmol/L;
5. hepatitis B virus resistance gene sequencing negative;
6. agree in the process of the study, do not participate in any other clinical studies or other anti HBV therapy;
7. before the beginning of the study, understand and sign the informed consent form approved by the ethics committee, and cooperate to conduct clinical research according to the requirements for the study.

Exclusion Criteria:

1. by the following evidences prompt suspected hepatocellular carcinoma: B ultrasound or imaging examination discover occupying lesion;B ultrasound normal but serum alpha fetoprotein (AFP) level has a continuous increasing trend; AFP > 100ng/ml, and after review, still so.
2. with liver disease acute exacerbation cause a transient liver function decompensation disease or baseline with clinical performance of decompensated liver disease;
3. serum creatinine ≥1.5mg/dl (≥130μmol/l);
4. the serum amylase > 2 times the normal reference upper limit value;
5. hemoglobin (male <100g/L, female <90g/L), white blood cell< 3.5* 109/L, platelet< 60 * 109/L;
6. combined with infection of HCV (anti -HCV positive), HIV, anti -HAV IgM positive, anti -HDV IgM positive, anti -HEV IgM positive, anti -EBV IgM positive, anti -CMV IgM positive, autoimmune hepatitis(such as the titer of anti nuclear antibody> 1:160) or activite liver disease caused by other known or unknown reason;
7. investigators consider that may interfere with the treatment,evaluation or compliance of the subjects, including any uncontrolled clinical significance of kidneys, heart, lungs, blood vessels, neurogenic, digestive system, metabolic diseases (diabetes, hyperthyroidism, adrenal disease), immune function disorder or tumor;
8. subjects with a history of alcoholism or drug abuse,investigators consider the subjects cannot comply with this protocol or affect the results analysis;
9. pregnancy,lactation or female subjects plan to conceive or the companions of male subjects plan to conceive during the study
10. 6 months before the study medication used immunosuppressants,immunomodulators(thymosin alpha), cytotoxic drugs;
11. 6 months before the study medication used anti HBV drug therapy (interferon, Lamivudine, Adefovir, Entecavir and Telbivudine, Tenofovir,etc);
12. plan or have had liver transplantation;
13. received other study drug treatment within 3 months prior to screening;
14. drug allergy history or allergic for Nucleoside or Nucleotide drug;
15. the subjects non compliance with the protocol or subjects exist any situation which investigators considered not suitable for participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
HBeAg serum conversion rate | Week 48
  The HBeAg serum conversion rate of the Test Group and the Control Group after 48 weeks treatment

SECONDARY OUTCOMES:
HBeAg serum conversion rate | Week 24, 72
  The HBeAg serum conversion rate of the Test Group and the Control Group for treatment week 24, week 72
HBeAg disappearance rate | Week 24, 48 and 72
  The HBeAg disappearance rate of the Test Group and the Control Group for treatment week 24, week 48 and week 72
HBV DNA titer | Week-4, 0,12,24,48,72 and 96
  The proportion of subjects for each observation point in HBV DNA titer decreased 2 logarithmic
The proportion of subjects for the HBV DNA can not be detected | Week 24, 48 and 72
  The proportion of subjects for the HBV DNA can not be detected in treatment week 24, week 48 and week 72
HBeAg and HBsAg titer | Week-4, 0,12,24,48,72 and 96
  The changes of HBeAg and HBsAg titer at each observation point
The quantitative changes of anti -HBc | Week-4, 0,12,24,48,72 and 96
  The quantitative changes of anti -HBc in each observation point
The variation of ALT | Week-4,24,48,72 and 96
  The variation of ALT in each observation point
The seroconversion rate of HBsAb and HBeAb | Week-4, 0,12,24,48,72 and 96
  The seroconversion rate of HBsAb and HBeAb in each observation point
The resistance mutation rate of HBsAb and HBeAb | Week-4, 0,12,24,48,72 and 96
  The resistance mutation ncidence of HBsAb and HBeAb in each observation point
The cumulative incidence of virologic breakthroughrate of HBsAb and HBeAb | Week-4, 0,12,24,48,72 and 96
  The cumulative incidence of virologic breakthroughrate of HBsAb and HBeAb in each observation point
The changes of relative immune parameters of the transfer factor in peripheral blood(the number of T lymphocytes and the expression levels of cytokines) | Week 0, 12, 24, 48, 72, 96
  The changes of relative immune parameters of the transfer factor in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Guiqiang Wang, Doctor, Study Chair — Peking University First Hospital; Maorong Wang, Doctor, Principal Investigator — China People's Liberation Army No. Eight One Hospital; Zheling Wang, Doctor, Principal Investigator — Qingdao Infectious Diseases Hospital; Zhiqiang zou, Doctor, Principal Investigator — Yantai Infectious Diseases Hospital; Peili Zhao, Doctor, Principal Investigator — The Third Hospital of Qinhuangdao City; Dexing Jia, Doctor, Principal Investigator — Weifang People's Hospital; Zhenghua Zhao, Doctor, Principal Investigator — Tai'an Central Hospital; Feng Gao, Doctor, Principal Investigator — Linyi People's Hospital; Sikui Wang, Doctor, Principal Investigator — Liaocheng People's Hospital; lingdao Huo, Doctor, Principal Investigator — The Third People's Hospital of Taiyuan; Yuping Ma, Doctor, Principal Investigator — Xi'an Eighth Hospital; Hongxu Zhang, Doctor, Principal Investigator — Luohe Central Hospital; Xu Zhang, Doctor, Principal Investigator — General Hospital of Ningxia Medical University